CLINICAL TRIAL: NCT05786014
Title: A Feasibility Study to Examine Two Remotely-monitored Exercise Interventions on Breast Cancer Patients Undergoing Cardiotoxic Chemotherapies
Brief Title: The Effects of Two Exercise Interventions on Breast Cancer Patients Undergoing Cardiotoxic Chemotherapies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Siddartha Angadi, Assistant Professor of Education, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 220287
Record Dates: First submitted 2023-03-13; First posted 2023-03-27 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Cardiotoxicity; Cardiovascular Diseases
Keywords: chemotherapy; cardiotoxicity; cardiorespiratory fitness
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity; Cardiovascular Diseases | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Subjects and investigators will not be blinded to treatment allocation. Outcome assessors will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate Intensity Walking (Experimental): Subjects allocated to moderate intensity walking will be given a gift card to purchase a paid of running shoes. A chest-based heart rate monitor and an activity tracker watch will be provided. Subjects will aim to achieve 150 minutes a week of moderate intensity walking. Subjects will also be receiving text messages, phone calls, and emails from study staff to gauge and encourage subject participation and physical activity.
  Interventions: Behavioral: Moderate Intensity Walking
- High Intensity Interval Exercise (Experimental): Subjects will receive a recumbent bike to be delivered and assembled to their home as well as a heart rate monitor and activity tracker. Subjects will undergo high intensity interval exercise 3 days a week, with the goal of achieving 85-90% of their heart rate max. Subjects will also be receiving text messages, phone calls, and emails from study staff to gauge and encourage subject participation and physical activity.
  Interventions: Behavioral: High Intensity Interval Exercise

INTERVENTIONS:
Behavioral: High Intensity Interval Exercise — Patients in the Cycling Intervention arm will undergo two training sessions at the exercise physiology core lab to ensure participants understand the intervention exercise protocol and can safely perform it at home. The Participants will perform high intensity interval training (HIIT) 3 days per week, with each session consisting of four, 4-min intervals at 85-90% peak heart rate (PHR), separated by 3 min at 50% PHR. Each training session will begin with a 10-minute warm-up at 50% of PHR and end with a 5-min cool down at 50% PHR. Subjects will then perform this exercise training at their own homes using recumbent exercise bikes provided by the investigators for that purpose. Study investigators will check in up to weekly with participants and remotely track exercise data and compliance via activity tracker.
  Arms: High Intensity Interval Exercise
Behavioral: Moderate Intensity Walking — Patients will undergo two familiarization training sessions in the exercise physiology core lab to ensure participants understands the walking intervention and can properly gauge intensity. Participants will be asked to walk briskly or jog so they achieve a moderate intensity (70-75% of the maximal heart rate achieved during the VO2peak test). The goal for participants in this condition will be to accumulate at least 150-minutes per week at this heart rate by brisk walking or jogging. Participants will also receive a gift card to be used to purchase a pair of walking shoes to facilitate their engagement.
  Arms: Moderate Intensity Walking

SUMMARY:
The purpose of this study is to determine if exercise preconditioning can mitigate the off target effects of chemotherapy treatment on measures of cardiovascular function, inflammatory responses, and quality of life.

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy affecting women in the US and survivors experience long-term health effects of chemotherapy. Exercise training is an efficacious treatment for preserving functional capacity and has shown promise in mitigating cardiac toxicity of breast cancer chemotherapy. However, supervised exercise is not a practical solution for all breast cancer survivors, as medically monitored exercise facilities are poorly dispersed in the US and poorly utilized by cancer patients. To improve reach of these programs, remotely monitoring exercise sessions may be necessary. However, effects of remotely-monitored exercise conditioning before and during adjuvant/neoadjuvant chemotherapy on cardiotoxic outcomes are unknown. Our study aims to address this gap by testing the feasibility of two types of remotely-monitored exercise interventions, an exercise bicycle intervention compared to a brisk walking intervention, in 20 UVA Breast Cancer Clinic patients undergoing cardiotoxic chemotherapies. Remotely-monitored exercise training will start one week prior to chemotherapy (preconditioning) and continue throughout adjuvant or neoadjuvant chemotherapy (which is typically 4 months in duration). Our multidisciplinary research team proposes four aims: 1) Determine the extent to which eligible patients can be successfully recruited, randomized, and retained; 2) Assess VO2peak, echocardiography derived left ventricular ejection fraction and left ventricular global longitudinal strain among these patients at baseline and at ~4 months; 3) Examine treatment engagement and intervention acceptability; and 4) Explore the relationship between engagement in the exercise training and psychosocial function.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or over
* diagnosis of breast cancer (Stage I-III or IV with minimal burden) and prescribed chemotherapy (TC (Docetaxel/Cyclophosphamide), AC (Doxorubicin/Cyclophosphamide followed by Paclitaxel), TCHP (Docetaxel, Carboplatin, Trastuzumab, Pertuzumab), TCH (Docetaxel/Carboplatin/Trastuzumab) with or without Pembrolizumab)
* Physician clearance for exercise training
* Speak/understand English

Exclusion Criteria:

* previous treatment with cardiotoxic chemotherapy
* medical/orthopedic comorbidities that preclude stationary cycling
* significant cardiac/renal/hepatic/hematological/pulmonary disease precluding exercise training
* unstable angina or myocardial infarction within 4-weeks prior to treatment
* complex ventricular arrhythmias or New York Heart Association class IV symptoms
* symptomatic severe aortic stenosis
* acute pulmonary embolus
* acute myocarditis
* History of untreated high-risk proliferative retinopathy
* History of retinal hemorrhage
* uncontrolled hypertension (systolic blood pressure > 180 mm Hg or diastolic blood pressure > 120 mm Hg)
* severe baseline electrolyte abnormalities
* medication non-compliance
* uncontrolled metabolic disease (diabetes with fasting blood sugar >300 mg/dl, thyrotoxicosis, myxedema)
* symptomatic peripheral vascular disease
* Pregnant women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
Subject Retention Percentage | 22 Weeks
  This is a feasibility study designed to determine the extent to which eligible patients can be successfully recruited, randomized, and retained. Endpoint data will be used to justify and provide point estimates for a fully powered study. Retention will be measured as a percentage of those enrolled who complete the study interventions.

SECONDARY OUTCOMES:
VO2peak | 22 Weeks
  Change in VO2peak (L/min) measured at pre-chemotherapy and post chemotherapy
Global Longitudinal Strain | 22 Weeks
  Global longitudinal strain (%) will be used to assess changes in cardiac contractile function and be measured by echocardiogram at pre-chemotherapy and post-chemotherapy
Ejection Fraction | 22 Weeks
  Ejection fraction (%) will be used to assess changes in cardiac contractile function and be measured by echocardiogram at pre-chemotherapy and post-chemotherapy
Diastolic Function | 22 Weeks
  E' and A' (cm/s) will be used to calculate the E'/A' ratio to assess for diastolic dysfunction and be measured by echocardiogram at pre-chemotherapy and post-chemotherapy
Brachial Artery Endothelium-Dependent Flow-Mediated Dilation | 22 Weeks
  Changes in endothelial function as measured by brachial artery endothelium-dependent flow-mediated dilation (%) at pre-chemotherapy and post-chemotherapy
Carotid-Femoral Pulse Wave Velocity | 22 Weeks
  Changes in arterial stiffness as measured by carotid-femoral pulse wave velocity (m/s) at pre-chemotherapy and post-chemotherapy
Blood pressure | 22 Weeks
  Brachial systolic and diastolic blood pressures (mmHg) will be measured at baseline and post-chemotherapy.
Lipid panels | 22 Weeks
  A lipid panel will be performed to measure total cholesterol, triglycerides, high-density lipoproteins, and low-density lipoprotein (mg/dl) to assess changes in cardiometabolic health at pre-chemotherapy and post-chemotherapy
Inflammation/Immune cell concentrations in peripheral circulation. | 22 Weeks
  Various markers of inflammation and immune cells will be measured at baseline, pre-chemo (following exercise pre-conditioning), midway through patient's prescribed treatment, and post-intervention to determine changes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia University Hospital, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No